CLINICAL TRIAL: NCT05571566
Title: The Impact of a Patient Education Tool on Parental Productivity and Anxiety: A Non-Randomized Control Trail
Brief Title: The Impact of a Patient Education Tool for Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sherif Emil, Professor of Pediatric Surgery, Surgery, and Pediatrics, McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-5195
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Appendicitis
Keywords: Parental Productivity; Parental Anxiety; Simple Appendicitis; Perforated Appendicitis; Patient Education Material; Appendicitis; Patient Survey; Parental Survey
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation phase (No Intervention): All patients with acute appendicitis who undergo appendectomies will be eligible to participate, and families will be consented prior to surgery. The explanation of the procedure will be done verbally by the surgeon as it is the standard care at the hospital. A parental anxiety assessment will be done before surgery with the Amsterdam Preoperative Anxiety and Information Scale (APAIS). In addition, an email from one of the primary caregivers will be collected, and the caregiver will receive an email with a link to the post-operative questionnaire 10 days post-discharge. At 14 days post-discharge, they will receive a reminder email again with the link to the questionnaire. All responses to the questionnaire are voluntary and anonymous.
- Post-implementation phase (Active Comparator): The education tool will be distributed to families whose child is undergoing an appendectomy. The explanation of the procedure will also be done verbally by the surgeon as it is the standard care at the hospital. The parental anxiety assessment will be done in the same way as above, before surgery with the Amsterdam Preoperative Anxiety and Information Scale (APAIS). In addition, the email of one of the primary caregivers will be collected, and the caregiver will receive an email with a link to the post-operative questionnaire 10 days post-discharge. At 14 days post-discharge, they will receive a reminder email with the link to the questionnaire. All responses to the questionnaire are voluntary and anonymous.
  Interventions: Other: Educational Book

INTERVENTIONS:
Other: Educational Book — An educational book with information about appendicitis for patients, parents and caregivers
  Arms: Post-implementation phase

SUMMARY:
Hypothesis/Study question (brief introduction of the question studied; about 5 lines)

Appendicitis is the most common acute surgical admission to the pediatric surgery service at the MCH. The need for surgery can provoke anxieties for patients. Patient education materials are meant to improve knowledge, set expectations, and improve the overall hospital experience for patients and their families, and are already being widely implemented for elective surgeries in the context of ERAS pathways. This study aims to develop an effective patient and family education tool, with the goal of improving patient education and satisfaction with care in the emergency surgery setting.

Study objectives

1. Utilize evidence-based methods to evaluate the success of implementation of a patient and family-centered education tool for appendicitis.
2. Develop and validate a pre- and post- education patient satisfaction and experience survey in the realm of pediatric surgery.
3. Inform the development of the education tool and survey through multidisciplinary and patient/family input.
4. Implement a patient/family-centered education tool in an emergency surgical setting.

DETAILED DESCRIPTION:
Methodology / Study design

1. Pilot phase Convenience sample of 10 patients diagnosed with acute appendicitis and their families will be selected to provide input on the patient and family experience survey tool. A convenience sample of 5 surgeons and 5 surgical nurses will also be solicited to provide feedback. The survey tool will be adapted based on the responses.
2. Pre-implementation phase All patients and their families with acute appendicitis who present to clinic for their routine follow-up appointment or are called for their phone-call follow up will be eligible to take a survey. All responses are voluntary and anonymous. The survey swill be available on an online platform so invited participants may conveniently participate in the study.
3. Post-implementation phase After the education pamphlet has been finalized and its distribution to families has begun, all patients and their families with simple or perforated appendicitis who had their initial presentation after the education pamphlet was available will be eligible to take a survey. All responses are voluntary and anonymous. The surveys will be available on an online platform so invited participants may conveniently and anonymously participate in the study.

Qualitative and descriptive statistics will be used to detect a difference in patient experience and satisfaction between the those who received the education tool and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregivers of all pediatric patients (0-17 years old) with acute appendicitis, including both perforated and non-perforated appendicitis cases, who have undergone an urgent appendectomy.

Exclusion Criteria:

* Patient or family does not understand English or French (education material available in only these two languages).
* Patient presenting for an elective interval appendectomy.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Parental Anxiety | 1 hour - during surgery
  Scores from the anxiety scale from both phases - adapted from Parental Anxiety Scale based on Amsterdam Preoperative Anxiety and Information Scale (APAIS) - 9 questions.
  The Parental Anxiety score is a Likert scale with 6 questions (each 1-5). The cutoff for anxiety is 13 points, anything over it is High anxiety.

SECONDARY OUTCOMES:
Parental Productivity | 10 & 14 days postoperatively
  Results from the online survey on parental productivity - adapted from Productivity and Disease Questionnaire (PRODISQ), the Health and Labor Questionnaire (HLQ) & additional literature. - 27 questions.
  The Parental Productivity survey will be a descriptive analysis and does not contain scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Emil, MD,CM, Principal Investigator — MUHC-RI
Locations (1):
- Research Institute of the McGill University Health Center/ Montreal Children's Hospital, Montreal, Quebec, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05571566/Prot_SAP_000.pdf